CLINICAL TRIAL: NCT04194866
Title: The Effect of Circadian Clock System on Perioperative Cognitive Function of Elderly Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Yanchao Yang, Principal investigator, Shengjing Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: circadian clock
Record Dates: First submitted 2019-12-10; First posted 2019-12-11 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Circadian Clock; Postoperative Cognitive Function; General Anesthesia; Elderly Patients
Keywords: circadian clock; postoperative cognitive function; general anesthesia; elderly patients

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Day group (Other): 60 patients scheduled for elective laparoscopic abdominal surgeries under general anesthesia were randomly assigned to receive operation in the Day Group ( 8:00-12:00)
  Interventions: Other: receiving operation during the day or at night
- Night group (Other): 60 patients scheduled for elective laparoscopic abdominal surgeries under general anesthesia were randomly assigned to receive operation in the Night Group (18:00-22:00)
  Interventions: Other: receiving operation during the day or at night

INTERVENTIONS:
Other: receiving operation during the day or at night — 120 patients scheduled for elective laparoscopic abdominal surgeries under general anesthesia were randomly assigned to receive operation in the Day Group (8:00-12:00) and in the Night Group (18:00-22:00)

SUMMARY:
Postoperative cognitive dysfunction (POCD) is a common postoperative complication in patients aged 65 and above. It refers to the cognitive function changes such as memory decline and attention loss after anesthesia and surgery. In serious cases, people may also experience personality changes and decline in social behavior ability, which will develop into irreversible cognitive impairment.Some studies reported that 25.8% of elderly patients presented POCD one week after non-cardiac surgery, and the incidence at 3 months after surgery was still 9.9%, which could increase the mortality in the first year after surgery.In recent years, studies have also proved that POCD is associated with patients' inability to perform their original jobs after non-cardiac surgery.Postoperative cognitive dysfunction seriously affects the clinical outcome, in addition to medical costs and other issues will bring an impact on the society and family.With the aging of the population, how to prevent cognitive dysfunction in elderly patients is a major challenge for perioperative management.There is a certain correlation between circadian rhythm and the dosage of general anesthesia, and postoperative sleep disturbance may be related to the effect of anesthesia and surgery on circadian rhythm.Preoperative sleep deprivation is known to be an independent risk factor for postoperative cognitive dysfunction (POCD), but the circadian mechanisms involved after general anesthesia are not yet clear

ELIGIBILITY:
Inclusion Criteria:

* preoperative sleep disorders
* did not receive any preoperative chemoradiotherapy
* the duration of surgery ≧3 hours

Exclusion Criteria:

* History of schizophrenia
* epilepsy
* parkinson's disease or myasthenia gravis
* Critical illness (preoperative American society of anesthesiologists (ASA) ASA >III)
* severe liver insufficiency (ChildePugh grade C)
* severe renal insufficiency (preoperative dialysis)
* neurosurgery

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
postoperative sleep quality of one night before surgery | one night before the surgery
  use sleep monitor to test the sleep quality one night before surgery
postoperative sleep quality of first night after surgery | the first night after surgery
  use sleep monitor to test the sleep quality first night after surgery
postoperative sleep quality of third night after surgery | the third night after surgery
  use sleep monitor to test the sleep quality third night after surgery

SECONDARY OUTCOMES:
Preoperative cognitive function test | one day before surgery
  use MMSE(Mini-mental state examination) scale to test the cognitive function one day before surgery. MMSE(Mini-mental state examination) is a simple test assessing several categories, such as orientation to time and place, short term memory, recall, attention, calculation, language and visuo-spatial abilities. Scores ranging from 30 to 24 usually indicate normal cognitive function, while lower scores suggest the presence of cognitive impairment: mild from 23 to 19, moderate from 18 to 10 and severe from 9 to 0
Postoperative cognitive function test of 6 weeks after surgery | 6 weeks after surgery
  use MMSE(Mini-mental state examination) scale to test the cognitive function 6 weeks after surgery. MMSE is a simple test assessing several categories, such as orientation to time and place, short term memory, recall, attention, calculation, language and visuo-spatial abilities. Scores ranging from 30 to 24 usually indicate normal cognitive function, while lower scores suggest the presence of cognitive impairment: mild from 23 to 19, moderate from 18 to 10 and severe from 9 to 0
Postoperative cognitive function test of 1 year after surgery | 1 year after surgery
  use MMSE(Mini-mental state examination) scale to test the cognitive function 1 year after surgery. MMSE(Mini-mental state examination) is a simple test assessing several categories, such as orientation to time and place, short term memory, recall, attention, calculation, language and visuo-spatial abilities. Scores ranging from 30 to 24 usually indicate normal cognitive function, while lower scores suggest the presence of cognitive impairment: mild from 23 to 19, moderate from 18 to 10 and severe from 9 to 0
Postoperative cognitive function test of 3 years after surgery | 3 years after surgery
  use MMSE(Mini-mental state examination) scale to test the cognitive function 3 years after surgery. MMSE(Mini-mental state examination) is a simple test assessing several categories, such as orientation to time and place, short term memory, recall, attention, calculation, language and visuo-spatial abilities. Scores ranging from 30 to 24 usually indicate normal cognitive function, while lower scores suggest the presence of cognitive impairment: mild from 23 to 19, moderate from 18 to 10 and severe from 9 to 0

CONTACTS AND LOCATIONS:
Overall Officials: Junchao Zhu, Study Director — Shengjing Hospital
Locations (1):
- Junchao hospital Zhu, Shenyang, Liaoning, China